CLINICAL TRIAL: NCT03926637
Title: Feasibility of the Multiple Sclerosis Performance Test for Assessment of Functional Performance Measures in Patients With Multiple Sclerosis
Brief Title: Feasibility of the Multiple Sclerosis Performance Test in Participants With Multiple Sclerosis
Status: Terminated | Type: Observational
Why Stopped: Biogen will stop any further development of the MSPT. The data collected thus far in the MSPT Feasibility Study allow us to answer the primary study objectives that are associated with assessing the feasibility of the MSPT in a clinical care setting.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-MSG-18-11424
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Multiple Sclerosis
Keywords: Clinically Isolated Syndrome
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Participants with MS, including CIS will complete the MSPT at their standard of care visits.
  Interventions: Other: Multiple Sclerosis Performance Test (MSPT)

INTERVENTIONS:
Other: Multiple Sclerosis Performance Test (MSPT) — Administered as specified in the treatment arm.

SUMMARY:
The primary objective is to evaluate the feasibility of the Multiple Sclerosis Performance Test (MSPT) in a clinical care setting when used by participants with Multiple Sclerosis (MS).

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with applicable participant privacy regulations
* Diagnosis of MS, including Clinically Isolated Syndrome
* Ability to understand the audio and visual instructions for the test modules
* Visual function, based on the investigator's clinical judgement that does not preclude an ability to interact with the Multiple Sclerosis Performance Test (MSPT).

Key Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Participants younger than 18 years of age, unless their parent or legal guardian provides the required signed and dated informed consent and authorization to use confidential health information and the participant provides assent in accordance with national and local subject privacy regulations

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a diagnosis of MS, including CIS will be offered study participation during their standard of care clinic visit or by contacting eligible participants identified from medical records.
Sampling Method: Non-Probability Sample
Enrollment: 3073 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Completing All Modules | Baseline to Month 24
Percentage of Participants Completing Each Individual Module | Baseline to Month 24
Percentage of Participants Skipping Modules | Baseline to Month 24
Average Time to Complete the Multiple Sclerosis Performance Test (MSPT) | Baseline to Month 24
Average Time to Complete Individual MSPT Modules | Baseline to Month 24
Frequency of Reasons for Not Completing MSPT Modules | Baseline to Month 24
Frequency Distribution of Demographic Characteristics of Participants Failing to Complete Specific MSPT Modules | Baseline to Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (32):
- United States (21):
  - Research Site, Berkeley, California
  - Research Site, Los Angeles, California
  - Research Site, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Owosso, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Teaneck, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Durham, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
- Research Site, Prague, Czechia
- Research Site, Strasbourg, France
- Italy (5):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Orbassano
  - Research Site, Roma
- Switzerland (2):
  - Research Site, Basel
  - Research Site, Bern
- United Kingdom (2):
  - Research Site, Camberley
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/